CLINICAL TRIAL: NCT00156507
Title: Improving Asthma Care for Very Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Halcyon Hill Foundation (Other)
Responsible Party: Jill S. Halterman, MD, MPH, Halcyon Hill Foundation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09653
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Parents of children in the experimental group receive asthma education prior to NICU discharge.
  Interventions: Behavioral: Asthma education for parents of very low birth weight infants

INTERVENTIONS:
Behavioral: Asthma education for parents of very low birth weight infants — Asthma education is provided to parents of children in the experimental group prior to nicu discharge.

SUMMARY:
Children born less than 1500 grams are being enrolled into a study to test the effectiveness of a parental educational intervention in reducing the risk of future breathing problems. The intervention teaches parents of these children how to reduce the risk of / and recognize breathing problems.

ELIGIBILITY:
Inclusion Criteria:

* Premature babies weighing less than 1500 grams at birth receiving care at Strong Memorial Hospital Neonatal Intensive Care Unit

Exclusion Criteria:

* Non-English speaking parents

Ages: 30 Days to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2003-01; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To evaluate whether education about asthma improves parent knowledge about the disease and its management and to evaluate whether education about asthma influences healthy behaviors to reduce breathing problems | 7-9 months post discharge

SECONDARY OUTCOMES:
To evaluate the feasibility of implementing the intervention in terms of cost and personnel time and to obtain parental feedback about the intervention. | 1-3 years post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jill S Halterman, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- Strong Memorial Hospital - Neonatal Intensive Care Unit, Rochester, New York, United States